CLINICAL TRIAL: NCT02079012
Title: Short- and Long-term Effects of a Walking Program ("Join the Walk?") on Physical Activity, Physical Fitness and Subjective Well-Being With Members of a Sports Federation for People With Mental Disorders (Psylos).
Brief Title: Effects of a Walking Program in People With Mental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Vlaamse Federatie voor Sport en Recreatie in de Geestelijke Gezondheidszorg (Unknown)
Responsible Party: Principal Investigator, Prof Filip Boen, Doctor, Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML10148
Record Dates: First submitted 2014-02-28; First posted 2014-03-05 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Mental Disorders
Keywords: Walking Program; Mental Disorders; Physical Activity; Physical Fitness; Anxiety; Depression; Self Determination
MeSH Terms: conditions — Mental Disorders; Motor Activity; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Receives:
  * An information session
  * A 10-week walking program (with documents, pedometer and three information sessions about motivation, a healthy diet and smoking cessation)
  * A physical activity diary (which also functions as a tool to check protocol-compliance)
  * Measurements
  Interventions: Behavioral: 10-week walking program
- Control group (No Intervention): Only receives measurements.

INTERVENTIONS:
Behavioral: 10-week walking program
  Arms: Intervention group

SUMMARY:
The purpose of this study is to investigate the short- and long-term effects of a 10-week walking program, based on the self-determination theory, in people with mental disorders. The investigators expect positive effects on:

* Physical fitness
* Physical activity
* Well-being (less feelings of anxiety, less feelings of depression) The investigators also expect underlying psychosocial processes to influence these effects.

DETAILED DESCRIPTION:
Framework: Previous research has shown beneficial health effects of a 10-week walking program in a senior organisation. Based upon the self-determination theory, similar results can be expected in people with mental disorders and could be highly relevant, given the fact that these people:

* Are often less active
* Have mental problems and often also comorbidities
* Are often socially isolated

Participants: Psylos tries to recruit a convenience sample of at least 100 participants for an intervention group (which will undertake the walking program) and 80 participants for a control group. All of them have to sign an informed consent. Due to attrition, at least 60 participants in the intervention group and 40 in the control group can be expected. A post hoc analysis, with detailed information about the variation in this population, may give additional information about the necessary power to obtain significant results.

Data analysis: First there will be examined whether the participants in both groups are equal at baseline according to relevant parameters (due to the non-randomisation). Second, to test the main effects, the difference scores will be examined between both groups. If certain assumptions are met, by an unpaired t-test; if not, by a non-parametric test. Finally (if relevant), the underlying psychosocial processes will be examined by regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Member of Psylos
* Medically approved by a physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in physical fitness pre - post | baseline, 10 weeks
  Via 6 minute walk test.
Change in physical fitness pre - follow-up | baseline, 6 months
  Via 6 minute walk test.
Change in physical activity pre - post | baseline, 10 weeks
  Via a questionnaire.
Change in physical activity pre - follow-up | baseline, 6 months
  Via a questionnaire.
Change in well-being pre - post | baseline, 10 weeks
  Via a questionnaire.
Change in well-being pre - follow-up | baseline, 6 months
  Via a questionnaire.

SECONDARY OUTCOMES:
Change in psychosocial parameters pre - post | baseline, 10 weeks
  Via a questionnaire.
Change in psychosocial parameters pre - follow-up | baseline, 6 months
  Via a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Boen, Prof., Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium